CLINICAL TRIAL: NCT01938989
Title: Effect of Blue Light Filtration on Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: A01311
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Cataract
Keywords: cataract; intraocular lens; IOL; blue light filter
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clear, then Blue Light Filter (Other): Clear clip-on glasses first, followed by blue light filter clip-on glasses, as worn over habitual correction
  Interventions: Device: Clear clip-on glasses; Device: Blue light filter clip-on glasses
- Blue Light Filter, then Clear (Other): Blue light filter clip-on glasses first, followed by clear clip-on glasses, as worn over habitual correction
  Interventions: Device: Clear clip-on glasses; Device: Blue light filter clip-on glasses

INTERVENTIONS:
Device: Clear clip-on glasses — Clip-on glasses with no light filtering properties
Device: Blue light filter clip-on glasses — Clip-on glasses with blue light filtering properties equivalent to AcrySof IOLs

SUMMARY:
The purpose of this study is to evaluate photostress recovery with blue light filter clip-on glasses among pseudophakes [ie, subjects in which the natural lens of the eye has been replaced with an artificial lens (intraocular lens) during cataract surgery]. This study will enroll subjects previously implanted with no blue light filter intraocular lenses (IOLs) for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery in both eyes with no blue light filtering intraocular lenses for at least 3 months;
* Good ocular health;
* 20/40 or better vision with best correction in both eyes;
* Willing to provide voluntary consent and sign informed consent form;
* Able to competently perform testing;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Ocular pathology, degeneration, or media opacity (cloudiness) that could impact study measurements;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefani Smith, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 study sites located in the US.
Pre-assignment Details: Of the 158 enrolled, 2 participants were exited as screen failures prior to randomization. This reporting group includes all randomized and treated participants (154). Note: 2 participants were randomized but not treated.
Period: Overall Study
Arm/Group | Clear, Then Blue Light Filter | Blue Light Filter, Then Clear
Started | 77 | 77
Completed | 77 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Overall: Blue light filter clip-on glasses and clear clip-on glasses worn over habitual correction in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 65

OUTCOME MEASURES:

1. Primary Outcome: Photostress Recovery Time
Description: Photostress Recovery Time is the time necessary to recover function (e.g., contrast discrimination) following exposure to a bright glare source. The subject fixated on an image (black and white grating) and underwent photostress (glare) for 5 seconds. Only 1 eye (study eye) was assessed.
Time Frame: Day 1
Population: This analysis population includes all participants with observation minus any major protocol deviations.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Blue Light Filter: Blue light filter clip-on glasses worn over habitual correction
- Clear: Clear clip-on glasses worn over habitual correction
Arm/Group | Blue Light Filter | Clear
Number analyzed (Participants) | 145 | 144
seconds | 5.66 (6.20) | 6.94 (7.16)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (30 Sep 2013 to 22 Jan 2014). This analysis group includes all enrolled participants.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. Reports of AEs were obtained through volunteered and elicited comments from the subjects.
Arm/Group | Blue Light Filter | Clear
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/158
Other Adverse Events (participants affected / at risk) | 0/158 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.